CLINICAL TRIAL: NCT07328464
Title: Occupational Exposure to Antineoplastic Drugs Among Physiotherapists in Healthcare Settings: From Assessing Internal Contamination to Implementing Co-constructed Prevention Measures
Brief Title: Occupational Exposure to Antineoplastic Drugs Among Physiotherapists in Healthcare Settings
Acronym: KINEMAC
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Collaborators: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: RCAPHM24_0277; 2025-A01689-40 (Other: AP-HM)
Record Dates: First submitted 2025-12-24; First posted 2026-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Internal and External Contamination of Physiotherapists by Antineoplastic Drugs
Keywords: Internal contamination; external contamination; physiotherapists; antineoplastic drugs; prevention measures; healthcare
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine samples collection and dermal wipe sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- physiotherapists: physiotherapists exposed to antineoplastic drugs in healthcare settings
  Interventions: Other: urine sample; Other: dermal wipe sampling; Other: questionnaires

INTERVENTIONS:
Other: urine sample — Internal contamination of antineoplastic drugs
Other: dermal wipe sampling — External contamination by antineoplastic drugs
Other: questionnaires — Participants will have questionnaires

SUMMARY:
Many antineoplastic drugs are considered "hazardous to handle" for healthcare professionals, notably because of their carcinogenic, mutagenic and/or reprotoxic effects. Occupational exposure occurs mainly through the cutaneous route, either by direct contact with the drug and/or indirectly through contact with treated patients and their excreta, or through contact with contaminated surfaces or textiles.

To date, physiotherapists have been little studied in terms of occupational exposure, even though they frequently perform care practices (massage, lymphatic drainage, limb mobilisation, respiratory physiotherapy) involving direct, prolonged and sustained skin contact with patients treated with antineoplastic drugs; these compounds may be eliminated in the sweat of the treated patient for several days after administration.

In this context, the present study aims to assess the occupational exposure of physiotherapists to antineoplastic drugs in healthcare settings. The primary objective is to estimate the prevalence of internal contamination of physiotherapists by antineoplastic drugs after performing one of the care practices (massage, lymphatic drainage, limb mobilisation, respiratory physiotherapy) selected for the study, in patients receiving intravenous treatment with antineoplastic drugs.

The secondary objectives are to describe for each antineoplastic drug studied the prevalence, the frequency of internal contamination of physiotherapists, and urinary concentration levels, to characterise the circumstances of exposure and the personal protective equipment worn, to describe the prevalence and the frequency of external cutaneous contamination on the hands and forearms of physiotherapists after performing an exposing care practice, to quantify this external cutaneous contamination, to identify the factors associated with internal and external contamination, and to co-develop preventive measures in collaboration with physiotherapists and stakeholders and to assess their acceptability.

This study is a non-interventional (RIPH3), cross-sectional and multicenter study conducted at AP-HM (Public Assistance for Marseille hospitals) and Bordeaux University Hospital (CHU de Bordeaux). Twenty physiotherapists will be included in this study. Internal contamination will be assessed over 100 observation visits and external contamination over 70 observation visits (all participants combined). Observation visit include at least one " an exposing care practice" (massage, lymphatic drainage, limb mobilisation, respiratory physiotherapy) performed on a patient who received an intravenous antineoplastic drug from a predefined list, within a time window of 4 to 72 hours after the start of injection.

- Internal contamination assessment (urine samples collection) For each observation visit, two urine samples of the physiotherapist participant will be collected: one sample within the 3 hours preceding the start of the work shift, and a second sample 6 to 10 hours after the end of the shift (or the next morning after waking up).

Data on exposure, activity and preventive practices (personal protective equipments worn) will be collected using an administered questionnaire (CRF). Information on the antineoplastic drugs administered to the patient receiving care by the physiotherapist will also be collected.

- Cutaneous external contamination assessment (dermal wipe sampling) For each observation visit, the physiotherapist will apply a standardized hands and forearms washing protocol, observed by the clinical research technician. Then, cutaneous swab samples will be taken immediately after the washing.

The physiotherapist will then perform an exposing care practice, limiting contact with the environment (e.g., door handles/surfaces), and new samples will be taken immediately after the exposing care practice, without prior decontamination of hands and forearms. A total of eight cutaneous swab samples (four before and four after an exposing care practice) will be collected per observation visit, according to a protocol validated by the reference laboratory.

The assessment of cutaneous external contamination of physiotherapists will be evaluated during visits separate from those used to study internal contamination.

The expected outcomes of this study are: an individual assessment of exposure and potential internal contamination and/or external dermal contamination, for each physiotherapist; traceability of exposure in occupational health medical records, for each physiotherapist; improved knowledge on the proportion of contaminated physiotherapists (prevalence and frequency) and knowledge on urinary and cutaneous concentration levels of antineoplastic drugs in physiotherapists; increased awareness among physiotherapists regarding these exposures; implementation of co-developed preventive actions aiming to reduce exposures to the lowest possible level; and improved professional practices and working conditions.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for individuals eligible for inclusion in the study:

Being a state-certified physiotherapist or hold an equivalent qualification, Working in one of the healthcare departments selected for the study, Being a man or woman aged 18 or over, Having received information about the study and not expressed any opposition to participating in it

Inclusion criteria for each physiotherapist observation visit as part of the internal contamination study:

Perform at least one physiotherapy treatment during this visit that must meet all of the following five criteria:

The physiotherapy treatment taken into account for this observation visit must be carried out in one of the healthcare departments selected for the study, This physiotherapy treatment being at least one of the following: massage and/or manual/lymphatic drainage and/or limb mobilisation and/or respiratory physiotherapy, This physiotherapy treatment being performed on a patient who has received intravenously at least one of the seven antineoplastic drugs studied, This physiotherapy treatment being performed within 4 to 72 hours of the start of intravenous administration of the antineoplastic drug(s) studied, This physiotherapy treatment is performed on a patient who is not in septic isolation and/or in a protected area.

Inclusion criteria for each physiotherapist observation visit as part of the external contamination study:

Perform at least one physiotherapy treatment during this visit that must meet all of the following five criteria:

The physiotherapy treatment taken into account for this observation visit, must be carried out in one of the healthcare departments selected for the study, This physiotherapy treatment being at least one of the following: massage and/or manual/lymphatic drainage and/or limb mobilisation and/or respiratory physiotherapy, This physiotherapy treatment being performed on a patient who has received intravenously at least one of the twelve antineoplastic drugs studied, This physiotherapy treatment being performed within 4 to 72 hours of the start of intravenous administration of the antineoplastic drug(s) studied, This physiotherapy treatment is performed on a patient who is not in septic isolation and/or in a protected area.

Exclusion Criteria:

Being a physiotherapy student, Being treated with one of the 12 antineoplastic drugs studied during the study or having been treated with one of them in the 2 months prior to the start of the study, Having a person and/or animal in their household who has been treated with one of the 12 antineoplastic drugs during the study or in the 2 months prior to the start of the study.

Physiotherapists who meet any of the following exclusion criteria for the observation visit will not be eligible for inclusion in the internal contamination assessment:

Being assessed for the internal contamination on the same day as the external contamination assessment, Being treated with one of the seven antineoplastic drugs studied during the study or having been treated with one of them during the two months preceding the observation visit, Having a person and/or animal in their household who is being treated with one of the seven antineoplastic drugs during the study or in the two months prior to the observation visit.

Exclusion criteria for each observation visit as part of the external contamination study

Physiotherapists who meet any of the following exclusion criteria for the studied physiotherapy treatment cannot be included in the external contamination assessment:

Being assessed for the external contamination on the same day as the internal contamination assessment, Performing this physiotherapy treatment while wearing a long-sleeved gown and/or long-sleeved overgown, Performing this physiotherapy treatment while using a cream and/or gel and/or oil, Being treated oneself with one of the 12 antineoplastic drugs studied during the study or having been treated with one of them during the 2 months preceding the physiotherapy treatment, Having a person and/or animal in their household who is being treated with one of the 12 antineoplastic drugs during the study or in the 2 months prior to the physiotherapy treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: physiotherapists in healthcare settings exposed to antineoplastic drugs
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Internal contamination (All antineoplastic drugs combined) | between month 0 and month 40 after inclusion
  The primary outcome measure is the assessment of the prevalence of internal contamination of physiotherapists by antineoplastic drugs based on urinary assays. Internal contamination corresponds to the presence of at least one of the seven antineoplastic drugs studied (cyclophosphamide, ifosfamide, etoposide, doxorubicin, daunorubicin, epirubicin, methotrexate), in at least one of the urine samples collected for each physiotherapist included.

SECONDARY OUTCOMES:
Internal contamination (for each antineoplastic drug studied) | between month 0 and month 40 after inclusion
  The secondary outcome measure is the prevalence and frequency of internal contamination by antineoplastic drugs among physiotherapists working in healthcare departments where patients are treated with these drugs
Urine concentration (for each antineoplastic drug studied) | between month 0 and month 40 after inclusion
  The secondary outcome measure is the urine concentration of the studied antineoplastic drugs, assaying by UHPLC-MS/MS.
External contamination | between month 0 and month 40 after inclusion
  The secondary outcome measure is the assessment of external contamination of physiotherapists by antineoplastic drugs based on cutaneous wiping sample. External contamination corresponds to the presence of at least one of the 12 antineoplastic drugs studied (cyclophosphamide, ifosfamide,étoposide, doxorubicine, daunorubicine, épirubicine, méthotrexate, paclitaxel, vincristine, pemetrexed, gemcitabine, dacarbazine), in at least one of the cutaneous wiping sample collected for each physiotherapist included.
Identification of factors associated with internal and external contamination | between month 0 and month 40 after inclusion
  Factors associated with internal contamination of physiotherapists will be studied based on data on exposure characteristics, on personal protective equipment use and urine sample results.
  Factors associated with external contamination of physiotherapists will be studied based on data on exposure characteristics, on personal protective equipment use and external contamination of physiotherapists.
Acceptability assessment of the co-constructed prevention measures | between month 35 and month 37 after inclusion
  The acceptability of these measures will then be assessed using a questionnaire during a semi-directive interview. The questionnaire will be constructed following the previous results. Time constraints and physical constraints related to physiotherapy practices such as massage and lymphatic drainage will be examined in particular

CONTACTS AND LOCATIONS:
Overall Officials: Francois Cremieux, Study Director — AP-HM
Locations (1):
- CHU de Bordeaux, Bordeaux, France